CLINICAL TRIAL: NCT03576586
Title: Improving Mental Health and Physiological Stress Responses in Mothers Following Traumatic Childbirth and in Their Infants: a Randomised Controlled Trial (START)
Brief Title: Swiss TrAumatic biRth Trial
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University of Lausanne (Other); University Hospital, Geneva (Other); University of Fribourg (Other); University of Zurich (Other)
Responsible Party: Principal Investigator, Antje Horsch, Assistant Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017-02142
Record Dates: First submitted 2018-06-04; First posted 2018-07-03 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Posttraumatic Stress Disorder; Acute Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic, Acute

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Brief computerized intervention (computer game "Tetris") plus usual care in the maternity department
  Interventions: Behavioral: Brief computerized intervention
- Control (Placebo Comparator): Attention placebo control (cognitive task for same amount of time) plus usual care in the maternity department
  Interventions: Behavioral: Attention placebo control

INTERVENTIONS:
Behavioral: Brief computerized intervention — Brief computerized intervention (computer game "Tetris") plus usual care in the maternity department
  Arms: Intervention
Behavioral: Attention placebo control — Brief cognitive task plus usual care in the maternity department
  Arms: Control

SUMMARY:
This randomized controlled study aims to investigate the effects of a brief computerized intervention (the computer game "Tetris") on intrusive memories and other posttraumatic stress symptoms following an emergency cesarean section (ECS). Women who have undergone an emergency cesarian section will be randomly allocated to either the brief computerized intervention plus usual care or an attention placebo control group plus usual care within the first 6 hours following the ECS. Women and their infants will be followed up at ≤ 1 week postpartum, 6 weeks postpartum, and 6 months postpartum. It is predicted that women given the brief computerized intervention will develop fewer intrusive memories and less posttraumatic stress symptoms than those who are not. This will inform the development of a simple computerized early intervention to prevent distressing psychological symptoms after a traumatic event, such as an ECS.

ELIGIBILITY:
Inclusion Criteria:

Women:

* had an ECS at ≥ 34 weeks gestation
* gave birth to a live baby
* answered with a score of ≥ 2 separately for at least two out of four screening questions regarding perceived threat
* gave written consent

Partners:

* if the woman agrees to participate
* was present at the childbirth
* gave written consent

Exclusion Criteria:

Women:

* don't speak French sufficiently well to participate in assessments
* have an established intellectual disability or psychotic illness
* severe illness of mother or infant (e.g. cancer, cardiovascular disease, severe neurodevelopmental difficulties, malformations)
* infant requires intensive care
* alcohol abuse and/or illegal drug use during pregnancy

Partner:

- don't speak French sufficiently well to participate in assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
presence and severity of PTSD symptoms: clinician-rated (mother) | 6 weeks postpartum
  Clinician-administered PTSD scale (CAPS): subscale and total scores
presence and severity of PTSD symptoms: self-report (mother) | 6 weeks postpartum
  PTSD Checklist (PCL-5): subscale and total scores

SECONDARY OUTCOMES:
frequency of intrusive traumatic memories (mother) | ≤ 1 week postpartum
  traumatic intrusions diary
presence and severity of ASD symptoms (mother) | < 6 hours after ECS, ≤ 1 week postpartum
  Acute Stress Disorder Scale (ASDS): subscale and total scores
presence and severity of PTSD symptoms: self-report (mother) | 6 months postpartum
  PTSD Checklist (PCL-5): subscale and total scores
presence and severity of PTSD symptoms: clinician-rated (mother) | 6 months postpartum
  Clinician-administered PTSD scale (CAPS): subscale and total scores
presence and severity of anxiety symptoms (mother) | < 6 hours after ECS, ≤ 1 week, 6 weeks, 6 months postpartum
  anxiety subscale of Hospital Anxiety and Depression Scale (HADS): subscale score
sleep time and duration (mother) | ≤ 1 week postpartum
  sleep diary
sleep quantity and quality (mother) | ≤ 1 week, 6 weeks, 6 months postpartum
  Pittsburgh Sleep Quality Index (PSQI): total score
presence and severity of depression symptoms (mother) | < 6 hours after ECS, ≤ 1 week, 6 weeks, 6 months postpartum
  Edinburgh Postnatal Depression Scale (EPDS): total score
sleep and physical activity (mother) | ≤ 1 week and 6 months postpartum
  Overnight accelerometer assessments
salivary cortisol: daily profile (mother and infant) | ≤ 1 week and 6 months postpartum
  daily profile
salivary cortisol: stress reactivity (mother and infant) | ≤ 1 week and 6 months postpartum
  stress reactivity
heart rate variability: resting state (mother and infant) | ≤ 1 week and 6 months postpartum
  resting state
heart rate variability: stress reactivity (mother and infant) | ≤ 1 week and 6 months postpartum
  stress reactivity
infant behavior (mother) | 6 months postpartum
  Infant Behavior Questionnaire-very short form: total and subscale scores
infant development | 6 months postpartum
  Bayley Scales of Infant Development (Bayley-III): clinician-rated
mother-infant-bonding (mother) | ≤ 1 week, 6 weeks, 6 months postpartum
  Mother-to-Infant-Bonding Scale (MIBS): total score
maternal emotional availability | 6 months postpartum
  Emotional Availability Scale: clinician-rated

OTHER OUTCOMES:
morningness-eveningness (mother) | ≤ 1 week postpartum
  Morningness-Eveningness Questionnaire (MEQ): total score
social support (mother, partner) | ≤ 1 week, 6 weeks, 6 months postpartum
  Modified Medical Outcomes Study Social Support Survey (MOS-8): total score
couple relationship adjustment (mother, partner) | ≤ 1 week, 6 weeks, 6 months postpartum
  Revised Dyadic Adjustment Scale (RDAS): subscale and total scores
parenting stress (mother, partner) | 6 months postpartum
  Parenting Stress Index - Short Form (PSI-SF): subscale and total scores
post-delivery perceived stress (mother) | ≤ 1 week postpartum
  Post-delivery Perceived Stress Inventory (PDPSI): subscale and total scores
postnatal perceived stress (mother) | 6 months postpartum
  Postnatal Perceived Stress Inventory (PPSI): subscale and total scores
self-reported life events (mother, partner) | ≤ 1 week and 6 months postpartum
  Life Events Questionnaire
breastfeeding | ≤ 1 week, 6 weeks, 6 months postpartum
  breastfeeding diary and questions
Dubowitz neurologic examination (infant) | ≤ 1 week postpartum
  structured clinical examination
frequency of intrusive traumatic memories (partner) | ≤ 1 week postpartum
  traumatic intrusions diary
presence and severity of PTSD symptoms: clinician-rated (partner) | 6 weeks, 6 months postpartum
  Clinician-administered PTSD scale (CAPS): subscale and total scores
presence and severity of PTSD symptoms: self-report (partner) | 6 weeks, 6 months postpartum
  PTSD Checklist (PCL-5): subscale and total scores
presence and severity of PTSD symptoms (partner) | ≤ 1 week postpartum
  Acute Stress Disorder Scale (ASDS): subscale and total scores
presence and severity of depression symptoms (partner) | ≤ 1 week, 6 weeks, 6 months postpartum
  Edinburgh Postnatal Depression Scale (EPDS): total scores
father-infant-bonding (partner) | ≤ 1 week, 6 weeks, 6 months postpartum
  Mother-to-Infant-Bonding Scale (MIBS): total score
participant feedback questionnaire (mother) | < 6 hours after ECS
  self-report questionnaire
treatment credibility/expectancy questionnaire (mother) | < 6 hours after ECS
  self-report questionnaire
presence and severity of anxiety symptoms (partner) | ≤ 1 week, 6 weeks, 6 months postpartum
  anxiety subscale of Hospital Anxiety and Depression Scale (HADS): subscale score
sleep quantity and quality (partner) | ≤ 1 week, 6 weeks, 6 months postpartum
  Pittsburgh Sleep Quality Index (PSQI): total score

CONTACTS AND LOCATIONS:
Overall Officials: Antje Horsch, D.Clin.Psych., Principal Investigator — University of Lausanne and Lausanne University Hospital
Locations (1):
- Prof. Antje Horsch, Lausanne, Switzerland

REFERENCES:
- [Background] Horsch A, Vial Y, Favrod C, Harari MM, Blackwell SE, Watson P, Iyadurai L, Bonsall MB, Holmes EA. Reducing intrusive traumatic memories after emergency caesarean section: A proof-of-principle randomized controlled study. Behav Res Ther. 2017 Jul;94:36-47. doi: 10.1016/j.brat.2017.03.018. Epub 2017 Apr 6. PMID 28453969
- [Derived] Deforges C, Sandoz V, Noel Y, Avignon V, Desseauve D, Bourdin J, Vial Y, Ayers S, Holmes EA, Epiney M, Horsch A. Single-session visuospatial task procedure to prevent childbirth-related posttraumatic stress disorder: a multicentre double-blind randomised controlled trial. Mol Psychiatry. 2023 Sep;28(9):3842-3850. doi: 10.1038/s41380-023-02275-w. Epub 2023 Sep 27. PMID 37759037
- [Derived] Sandoz V, Deforges C, Stuijfzand S, Epiney M, Vial Y, Sekarski N, Messerli-Burgy N, Ehlert U, Bickle-Graz M, Morisod Harari M, Porcheret K, Schechter DS, Ayers S, Holmes EA, Horsch A; START Research Consortium. Improving mental health and physiological stress responses in mothers following traumatic childbirth and in their infants: study protocol for the Swiss TrAumatic biRth Trial (START). BMJ Open. 2019 Dec 30;9(12):e032469. doi: 10.1136/bmjopen-2019-032469. PMID 31892657